CLINICAL TRIAL: NCT00312299
Title: Posterior Capsule Opacification After Implantation of Square Edge PMMA, Round Edge PMMA and Acrysof Intraocular Lenses: Randomized Controlled Study
Brief Title: Posterior Capsule Opacification Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2PR1210608
Record Dates: First submitted 2006-04-07; First posted 2006-04-10 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Cataract
Keywords: Double-Blind Method; Clinical Trials, Randomized; Lenses, Intraocular; Prospective Studies; PMMA; Visual acuity
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 A - Square edge PMMA IOL (Experimental): 50 patientes will recieve square edge PMMA IOL
  Interventions: Device: Square edge PMMA IOL
- 1B (Active Comparator): In group 1, 50 eyes will receive round edge PMMA IOL
  Interventions: Device: Round edge PMMA IOL
- 2A (Experimental): In group 2, 50 eyes will receive square edge PMMA IOL
  Interventions: Device: Square Edge PMMA IOL
- 2B (Active Comparator): In group 2, 50 eyes will receive acrysof IOL
  Interventions: Device: Acrysof IOL

INTERVENTIONS:
Device: Square edge PMMA IOL — Arm 1 A - Square edge PMMA IOL
  Other Names: TrueEdge IOL; S3602SQ
  Arms: Arm 1 A - Square edge PMMA IOL
Device: Round edge PMMA IOL — Round edge PMMA IOL
  Other Names: S3602
  Arms: 1B
Device: Acrysof IOL — Acrysof IOL
  Other Names: SA60AT
  Arms: 2B
Device: square Edge PMMA IOL — Square edge PMMA intra ocular lens
  Arms: Arm 1 A - Square edge PMMA IOL
Device: Square Edge PMMA IOL — Square Edge PMMA IOL lens
  Arms: 2A

SUMMARY:
First object is to compare square edge PMMA with round edge PMMA IOL where the materials are same. Next objective is to compare square edge PMMA IOL with Acrysof IOL where the materials are different

DETAILED DESCRIPTION:
Cataract is the vision impairing disease characterized by gradual, progressive thickening of the lens. Posterior Capsular Opacification (PCO) remains the most frequent long term complication. This is initiated by the migration and proliferation of residual lens epithelial cells from the lens equator in the space between the posterior capsule and intraocular lens (IOL)

The combination of IOL material and a sharp edged design is effective in preventing PCO. Aurolab has developed 360 degree square edge IOL with polymethyl methacrylate (PMMA)

100 bilateral senile cataract patients are going to be recruited. First group of 50 patients will receive square edge PMMA in one eye and round edge PMMA in fellow eye. Another group of 50 patients will receive square edge PMMA in one eye and acrysof in fellow eye. PCO will be assessed during each follow up using EPCO software.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 65 years
* Bilateral senile cataract
* Pupil should be at least 7mm dilated
* Nuclear sclerosis grade I, II and III
* Patient willing for second eye surgery within 3 months

Exclusion Criteria:

* Debilitated old patients
* Cardiac and serious illness
* Intraoperative complications including PC rent, Zonular dialysis and Rhexis tear
* Inherent zonular weakness
* Glaucoma patients
* Relative afferent papillary defect (RAPD)
* Shallow anterior chamber
* Pseudoexfoliation
* Traumatic cataract
* Uveitis and complicated cataract
* One eyed patients
* Corneal pathology
* Post segment pathology including diabetic retinopathy
* Dense Posterior subcapsular cataract (PSCC) and Posterior polar cataract (PPC)
* High myopic and hyperopic patient

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-04; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
PCO | 1 Day, 1 Month, 6 Month, 1 Year, 2 Year, 3 Year, 4 Year, 5 Year

SECONDARY OUTCOMES:
Visual Acuity | 1 Day, 1 Month, 6 Month, 1 Year, 2 Year, 3 Year, 4 Year, 5 Year

CONTACTS AND LOCATIONS:
Overall Officials: Haripriya Aravind, MBBS, MS, Principal Investigator — Aravind Eye Hospital, Madurai
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India